CLINICAL TRIAL: NCT00109252
Title: An Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of 1.0 mg/kg Subcutaneously Administered Efalizumab Followed by Efalizumab Taper in Adults With Plaque Psoriasis Previously Enrolled in Study ACD2390g
Brief Title: A Study to Evaluate Raptiva in Adults With Plaque Psoriasis Previously Enrolled in Study ACD2390g
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACD2391g
Record Dates: First submitted 2005-04-26; First posted 2005-04-26 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; Topical
MeSH Terms: conditions — Psoriasis | interventions — efalizumab

INTERVENTIONS:
Drug: Raptiva (efalizumab)

SUMMARY:
This is an open-label, multicenter study designed to evaluate the efficacy and safety of efalizumab administered at weekly SC (subcutaneous) doses of 1.0 mg/kg followed by efalizumab taper in subjects with plaque psoriasis who previously participated in Study ACD2390g.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Previous participation in Study ACD2390g
* For women of childbearing potential, continued use of an acceptable method of contraception for the duration of their participation in the study
* Willingness to continue to hold sun exposure reasonably constant and to avoid use of tanning booths or other UV light sources throughout the study

Exclusion Criteria:

* Any medical condition that, in the judgment of the investigator, would jeopardize the subject's safety following exposure to efalizumab
* Systemic therapy for psoriasis (ET Day 0 through FU Day 84 or upon relapse or unusual presentation of psoriasis in the FU period, whichever occurs first)
* Systemic immunosuppressive drugs for other indications (ET Day 0 through FU Day 84)
* Topical therapies for psoriasis (ET Day 0 through ET Day 84)
* Live virus or bacteria vaccines (ET Day 0 through FU Day 84)
* Other vaccines or allergy desensitization (it is recommended that these be scheduled after FU Day 84)
* Other experimental drugs or treatments (ET Day 0 through FU Day 84)
* Beta-Blockers, ACE inhibitors, interferons, quinidine, antimalarial drugs, or lithium (if clinically indicated, such medications are allowed but the dosage should be held constant between ET Day 0 and TT Day 84)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 2002-01; Study Completion 2003-04 (Actual)